CLINICAL TRIAL: NCT04282226
Title: Randomised Cross-over Study of the Effect of Transcutaneous Vagal Nerve Stimulation (tVNS) on Brain Activation at Rest and During Oesophageal Pain in Healthy Humans
Brief Title: Brain Effect of Vagal Nerve Stimulation at Rest and Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There was a serious delay in the study due to the COVID pandemic. So the grant period was over.
Sponsor: Queen Mary University of London (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: QMERC2017/59
Record Dates: First submitted 2020-02-14; First posted 2020-02-24 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteer
Keywords: transcutaneous vagal nerve stimulation; functional magnetic resonance imaging; visceral pain; oesophageal stimulation
MeSH Terms: conditions — Visceral Pain

STUDY DESIGN:
Intervention Model Description: Randomised, cross-over design with placebo control
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tVNS (Active Comparator): The tVNS device will be attached to the left aspect of the neck to stimulate the cervical branch of the vagal nerve and connected to an MR safe electrical
  Interventions: Device: active transcutaneous Vagal Nerve Stimulation (tVNS)
- sham tVNS (Placebo Comparator): The tVNS device will be attached to anatomically distinct from the cervical branch of the vagal nerve.
  Interventions: Device: sham transcutaneous Vagal Nerve Stimulation (tVNS)

INTERVENTIONS:
Device: active transcutaneous Vagal Nerve Stimulation (tVNS) — The tVNS device will be attached to the left aspect of the neck to stimulate the cervical branch of the vagal nerve and connected to an MR safe electrical stimulator.
  Arms: active tVNS
Device: sham transcutaneous Vagal Nerve Stimulation (tVNS) — The tVNS device will be attached to anatomically distinct from the cervical branch of the vagal nerve.
  Arms: sham tVNS

SUMMARY:
Pain is a ubiquitous distressing sensory experience and is the most frequent symptom in numerous gastrointestinal disorders including inflammatory bowel disease (IBD) and irritable bowel syndrome (IBS). Visceral pain is especially difficult to treat with conventional medications and new treatments are needed.

Recently, the relationship between autonomic nerve system (ANS) and pain has gathered attention because it could represent an effective treatment target for visceral pain. The parasympathetic nervous system (PNS), one of the two main branches of the ANS, is considered to play an important role for analgesia possibly due to vagal nerve-mediated activation of key brain areas implicated in descending analgesia of pain. Transcutaneous vagal nerve stimulation (tVNS) can non-invasively modulate vagal nerve and be expected as a new method to treat visceral pain. For example, the preliminary study showed that vagal nerve stimulation experimentally modulated cardiac vagal tone (CVT) and prevented the development of acid-induced oesophageal hyperalgesia.

Disturbances in ANS function have been reported not only in IBS patients but also in fibromyalgia and chronic pelvic pain syndrome. Many of these disorders have been associated with differences in brain structure and/or function as demonstrated by the use of structural and functional magnetic resonance imaging (fMRI). Of note, the investigators have recently shown that these differences in brain structure and function may be in part attributable to the aforementioned disturbance in ANS function, adding weight to the proposition that autonomic neuromodulation may be efficacious in pain disorders. For instance, in healthy participants the investigators have recently shown, using functional connectivity analysis, that higher resting parasympathetic CVT predicts the engagement of a subcortical functional network that is implicated in descending analgesia, thereby supporting the notion that vagal-mediated analgesia is achieved via descending inhibitory pathways1,4. Thus, tVNS seems a reasonable method to treat pain. However, to date, the precise real-time effect of tVNS on brain function, including during the processing of visceral pain is unknown.

Hence, the aims of this study are to investigate the real-time effect of tVNS compared to sham stimulus on brain activity whilst experiencing acute oesophageal pain, using fMRI in double-blind, randomised crossover study of tVNS vs sham stimulation in healthy subjects.

DETAILED DESCRIPTION:
Following informed written consent and screening questionnaires to characterize psychophysiological traits including personality and anxiety/depression inventory, each subject will have a nasogastric tube inserted with the attached distensible balloon positioned in the distal oesophagus. Painful oesophageal stimulation will be achieved by inflation of the balloon to a pain threshold pre-determined in each subject, defined as the point at which subject describes the transition from sensation to pain. The MR-safe tVNS probe will be attached to the neck for cervical vagal nerve-directed tVNS, and subjects will then be positioned in the MRI scanner. Real-time activity of the ANS will be monitored by heart rate variability as described in the previous study, which has been adapted for use in the MR-environment. All subjects will undergo MRI. For each visit, there will be two scanning periods. High-resolution structural imaging will first be required, and subsequently resting fMRI data will be acquired whilst subjects are asked to relax in the scanner, and their baseline autonomic tone is monitored, using validated methods of acquiring ANS data. This will illustrate a brain signature of real-time brain activity mapped to their parasympathetic tone.

Subjects will then be randomised to either the active-tVNS paradigm or sham and a second fMRI data acquisition will then be performed so as to acquire brain activity in conjunction with active and sham-tVNS. Following this, painful oesophageal stimulation will be repeated 20 times while active or sham tVNS continues. Following a two-week washout period, subjects will be crossed over and re-examined to receive the intervention they did not receive in visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants (defined as those without pre-existing medical comorbidity) from staff, students and the local population of Queen Mary, University of London and/or King's College London
* Inclusion will be determined on the basis of availability. They should be able to attend the Denmark Hill King's College London Campus for 2 sessions.
* Women should be studied in the follicular phase of their menstrual cycle or taking oral contraceptives.

Exclusion Criteria:

* Participants unable to provide informed consent
* Participants with any systemic disease or medications that may influence the autonomic nervous system (e.g. beta-agonists or Parkinson's disease)
* Pregnant or breastfeeding females
* Participants unable to lie flat in the MRI scanner, suffer from claustrophobia or are unsuitable for MRI scanning due to contraindications, comorbidity or in situ metalwork
* Current smokers
* History of anxiety or depression, or hospital anxiety or depression score >8
* History of drug or alcohol abuse
* Patients who have cardiovascular condition problems
* Patient with cochlear implants
* Recent nasal trauma, base of skull fracture and/or facial surgery that would contraindicate insertion of a nasogastric tube
* A positive urinary drugs screen
* Head circumference exceeding the limits of the scanner
* Not meeting any of the inclusion criteria above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The effect of tVNS compared to sham stimulus on brain activity whilst experiencing oesophageal pain | 2 weeks
  Comparison of fMRI results between sham and active tVNS.

SECONDARY OUTCOMES:
The effect of tVNS on functional brain activity at baseline and following painful oesophageal stimulation | 2 weeks
  Comparison of fMRI results before and after oesophageal stimulation.
The effect of tVNS on participant pain ratings to acute oesophageal pain | 2 weeks
  Participants is asked to rate the severity of the pain they received using a simple 100-point visual analogue scale. (The minimum and maximum values are 1 and 100, respectively)
The effect of baseline autonomic tone on structural brain morphology (both gray and white matter) | 2 weeks
  Cardiac vagal tone is calculated using electrocardiogram data to evaluate autonomic tone, which is measured on a linear vagal scale (LVS). The correlation between cardiac vagal tone and MRI results is evaluated.
The effect of tVNS on resting brain function coupled to resting parasympathetic tone, compared to sham stimulus | 2 weeks
  fMRI results are compared between active and sham tVNS.
The correlation of structural MR, DTI and resting fMRI data on the efficacy of tVNS for use in visceral pain | 2 weeks
  Investigating whether or not brain morphology predict efficacy with tVNS in pain.
The effect of tVNS on state anxiety following oesophageal pain. | 2 weeks
  State and Trait Anxiety Inventory state, trait (Maximum and minimum values are 80 and 20, respectively. The higher value indicates more nervous status) is used.

CONTACTS AND LOCATIONS:
Overall Officials: Qasim Aziz, Study Chair — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No